CLINICAL TRIAL: NCT01430468
Title: Comparison of Glenoid Component Position Using Patient Specific Instruments Versus Standard Surgical Instruments: A Randomized Prospective Clinical Trial
Brief Title: Patient Specific Instruments Versus Standard Surgical Instruments
Acronym: TIOSO-GPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Joseph Iannotti, Institute Chairman, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CCF 10-582; TECH 09-073 (Other Grant/Funding Number: State of Ohio BRCP research grant)
Record Dates: First submitted 2011-09-01; First posted 2011-09-08 (Estimated); Results first posted 2017-03-07 (Actual); Last update posted 2020-06-01 (Actual); Status verified 2020-01

CONDITIONS: Total Shoulder Arthroplasty
Keywords: Glenoid component position; patient specific instruments

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Glenoid Positioning System (Experimental): For the patients randomized to the GPS group, the surgeon will be given the GPS patient specific instrumentation and a model of the glenoid surface showing the exact placement and fit of the GPS alignment instruments.
  Interventions: Procedure: Glenoid Positioning System
- Standard Group (No Intervention): Each surgeon will use their standard methods of pre-operative planning using the pre-operative x-rays and CT scan.

INTERVENTIONS:
Procedure: Glenoid Positioning System — Design and fabrication of patient specific instrument for placement of a guide pin to be used to aid in bone preparation for placement of a metaglene and its fixation screws or anatomic glenoid component
  Arms: Glenoid Positioning System

SUMMARY:
Comparison of Glenoid Component Position Using Patient Specific Instruments Versus Standard Surgical Instruments: A Randomized Prospective Clinical Trial

DETAILED DESCRIPTION:
This is a non blinded prospective randomized clinical trial to define the efficacy of a new technology developed at the Cleveland Clinic to improve the positioning of the glenoid component in total shoulder arthroplasty. The Cleveland Clinic research team has worked on the development and validation of this new technology for the last six years. The investigators have validated the pre-operative planning software and published the results in the peer review literature (1, 7, 8, 9). The investigators have used this software in the planning of total shoulder surgery over the last three years. The investigators have validated the accuracy and reproducibility of the patient-specific instrumentation in both cadaver shoulders and Sawbones models of the shoulder using multiple surgeons. These studies also validated our ability to precisely measure component position using 3D CT scan imaging after placement of the implants in a pre-clinical cadaver study, thereby validating our ability to accurately measure and compare component position between the groups described in this proposed clinical trial. The investigators have also proven the ability of the software and techniques to produce an accurate representation of the glenoid morphology in patients with osteoarthritis or rotator cuff deficient arthritis in 13 patients. This was an IRB approved patient safety study performed at the Cleveland Clinic. The investigators have performed extensive studies of the materials and processes for the fabrication, sterilization and packaging of the patient specific instruments. The investigators have selected materials and processes that have met all of the FDA requirements for use of these materials and processes as clinical devices in vivo. These devices (non implanted instruments) are generally classified by FDA as a Class I device not having significant clinical risk. The investigators have studied the materials and process to produce accurate instruments that meet the clinical specification for fit onto the surrogate glenoid surfaces and maintain this shape and fit after sterilization. These same patient specific instruments have been tested in pre-clinical trials (Sawbones and Cadavers), demonstrating their ability to perform the functions specified with a high level of accuracy and much better than the use of standard generic instruments.

ELIGIBILITY:
Inclusion Criteria:

* All patients otherwise indicated for primary reverse or anatomic total shoulder replacement that are able to get a pre-operative CT scan at the Cleveland Clinic will be considered eligible for enrollment. All patients will be consented in the office as part of the pre-operative consent for surgery and all will need to randomization at the time of surgery

Exclusion Criteria:

* Patients will be excluded if they have significant metal in the joint that results in metal artifact on the CT scan, thereby compromising the ability to visualize the glenoid on the pre-operative simulator.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2010-09; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph P. Iannotti, MD, PhD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD with other researchers.

REFERENCES:
- [Background] Codsi MJ, Bennetts C, Gordiev K, Boeck DM, Kwon Y, Brems J, Powell K, Iannotti JP. Normal glenoid vault anatomy and validation of a novel glenoid implant shape. J Shoulder Elbow Surg. 2008 May-Jun;17(3):471-8. doi: 10.1016/j.jse.2007.08.010. Epub 2008 Mar 7. PMID 18328741
- [Background] Matsen FA 3rd, Clinton J, Lynch J, Bertelsen A, Richardson ML. Glenoid component failure in total shoulder arthroplasty. J Bone Joint Surg Am. 2008 Apr;90(4):885-96. doi: 10.2106/JBJS.G.01263. PMID 18381328
- [Background] Franta AK, Lenters TR, Mounce D, Neradilek B, Matsen FA 3rd. The complex characteristics of 282 unsatisfactory shoulder arthroplasties. J Shoulder Elbow Surg. 2007 Sep-Oct;16(5):555-62. doi: 10.1016/j.jse.2006.11.004. Epub 2007 May 16. PMID 17509905
- [Background] Gutierrez S, Comiskey CA 4th, Luo ZP, Pupello DR, Frankle MA. Range of impingement-free abduction and adduction deficit after reverse shoulder arthroplasty. Hierarchy of surgical and implant-design-related factors. J Bone Joint Surg Am. 2008 Dec;90(12):2606-15. doi: 10.2106/JBJS.H.00012. PMID 19047705
- [Background] Hafez MA, Chelule KL, Seedhom BB, Sherman KP. Computer-assisted total knee arthroplasty using patient-specific templating. Clin Orthop Relat Res. 2006 Mar;444:184-92. doi: 10.1097/01.blo.0000201148.06454.ef. PMID 16446589
- [Background] Iannotti JP, Spencer EE, Winter U, Deffenbaugh D, Williams G. Prosthetic positioning in total shoulder arthroplasty. J Shoulder Elbow Surg. 2005 Jan-Feb;14(1 Suppl S):111S-121S. doi: 10.1016/j.jse.2004.09.026. PMID 15726070
- [Background] Scalise JJ, Bryan J, Polster J, Brems JJ, Iannotti JP. Quantitative analysis of glenoid bone loss in osteoarthritis using three-dimensional computed tomography scans. J Shoulder Elbow Surg. 2008 Mar-Apr;17(2):328-35. doi: 10.1016/j.jse.2007.07.013. Epub 2008 Jan 22. PMID 18218326
- [Background] Scalise JJ, Codsi MJ, Bryan J, Brems JJ, Iannotti JP. The influence of three-dimensional computed tomography images of the shoulder in preoperative planning for total shoulder arthroplasty. J Bone Joint Surg Am. 2008 Nov;90(11):2438-45. doi: 10.2106/JBJS.G.01341. PMID 18978413
- [Background] Scalise JJ, Codsi MJ, Bryan J, Iannotti JP. The three-dimensional glenoid vault model can estimate normal glenoid version in osteoarthritis. J Shoulder Elbow Surg. 2008 May-Jun;17(3):487-91. doi: 10.1016/j.jse.2007.09.006. Epub 2008 Feb 20. PMID 18282721

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Glenoid Positioning System | Standard Group
Started | 22 | 22
Completed | 15 | 16
Not Completed | 7 | 6
Not completed — Physician Decision | 2 | 1
Not completed — Withdrawal by Subject | 5 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Glenoid Positioning System | Standard Group | Total
Number analyzed (Participants) | 15 | 16 | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.1 (6.8) | 67.3 (9.5) | 68.2 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 11 | 19
  Male | 7 | 5 | 12
Region of Enrollment [Number; unit: participants]
  United States | 15 | 16 | 31
Pre-operative retroversion [Mean (Standard Deviation); unit: Degrees] — Degrees of retroversion from 3-D CT scan
  Degrees | -14.8 (10.1) | -11.3 (13.3) | -13.0 (11.8)

OUTCOME MEASURES:

1. Primary Outcome: Comparing Glenoid Component Positioning to Pre Operative Planning
Description: Final implant position will be determined by comparing the position of the glenoid component on the post-operative CT scans with the implant position planned pre-operatively on the surgical simulator. These measurements will be in degrees.
Time Frame: 1 month post op
Measure: Mean (Standard Deviation); unit: Degrees
Arm/Group | Glenoid Positioning System | Standard Group
Number analyzed (Participants) | 15 | 16
Degrees | 4.3 (4.5) | 6.9 (4.4)
Statistical Analysis 1: Comparison: Glenoid Positioning System vs Standard Group; The absolute difference between the actual outcome and the planned outcome was compared between the standard surgical group and the glenoid positioning system group with use of a Student t test. Results were considered to be significant at p < 0.05; Test type: Equivalence — With use of previously established criteria for a malpositioned glenoid, deviations of greater than 10 degrees of version from the planned placement were considered relevant; p = 0.11, t-test, 2 sided — P-value was calculated. Threshold for statistical significance (p<0.05)

2. Secondary Outcome: Intra-operative Photographs
Description: Intra-operative photographs will be used to qualitatively, not quantitatively, to document the surgical steps and may be useful to explain a deviation in the surgery than what would have been expected by the pre-operative simulator. No quantitative data will be collected from the photographs.
Time Frame: Intra-operative
Population: Number participants with deviation in the surgery than expected by the pre-operative simulator.
Measure: Count of Participants; unit: Participants
Arm/Group | Glenoid Positioning System | Standard Group
Number analyzed (Participants) | 15 | 16
Participants | 0 | 0

ADVERSE EVENTS:
Arm/Group | Glenoid Positioning System | Standard Group
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/16
Other Adverse Events (participants affected / at risk) | 0/15 | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes